CLINICAL TRIAL: NCT05249517
Title: Telerehabilitation Based Pain Neuroscience Education on Patients With Non-specific Chronic Neck Pain: A Double-Blinded Randomized Controlled Trial
Brief Title: Telerehabilitation Based Pain Neuroscience Education on Patients With Non-specific Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ahmet Ozturk, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DokuzEU_AO
Record Dates: First submitted 2022-01-12; First posted 2022-02-21 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Neck Pain
Keywords: Neck pain; Telerehabilitation; Pain neuroscience education
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education (PNE) (Experimental): Telerehabilitation based pain neuroscience education
  Interventions: Other: Pain Neuroscience Education
- Exercise + PNE (Active Comparator): Telerehabilitation based progressive submaximal exercise program and PNE
  Interventions: Other: Progressive submaximal exercise program

INTERVENTIONS:
Other: Pain Neuroscience Education — Pain Neuroscience Education (PNE) is a patient education approach that explains in detail the neurobiology, neurophysiology of pain, and the processing of pain by the nervous system in the management of chronic pain.
  Arms: Pain Neuroscience Education (PNE)
Other: Progressive submaximal exercise program — It has been shown that the long-term results of the use of PNE in addition to physiotherapy are more effective in reducing pain and disability. It has been reported that progressive submaximal exercise program including cervicothoracic strengthening, endurance, flexibility, and coordination exercises has positive effects on chronic neck pain, related disability, quality of life and mood.
  Arms: Exercise + PNE

SUMMARY:
In this study, the effects of 6-week telerehabilitation-based Pain Neuroscience Education and exercise training in participants with Non-specific Chronic Neck Pain will be investigated.

DETAILED DESCRIPTION:
Neck pain is a general health problem that is very common in society and affects daily life activities by causing disability. Non-specific chronic neck pain is defined as "continuous neck pain that persists for 12 weeks or longer beyond the healing process without any known specific pathology. Chronic pain is considered to be a complex problem in which cognitive and emotional factors, as well as biological factors, significantly affect the perception of pain. In the last decade, a patient education model that educates people about the neurobiology and neurophysiology of pain has been recognized as an intriguing approach to the management of chronic pain. Pain Neuroscience Education (PNE) is a patient education approach that explains in detail the neurobiology, neurophysiology of pain, and the processing of pain by the nervous system in the management of chronic pain. In the literature, there is evidence supporting the use of PNE in reducing pain and disability and overcoming the psychosocial factors of chronic pain.

While the Covid-19 pandemic has made telerehabilitation applications widespread, it has also shown us its necessity, but until now, no study in which Pain Neuroscience Education was carried out with the telerehabilitation method has been found in the literature.

This study aimed to perform Pain Neuroscience Education with the telerehabilitation method on patients with non-specific chronic neck pain and to examine the effects on pain-related factors, disability, and quality of life.

It has been shown that the long-term results of the use of PNE in addition to physiotherapy are more effective in reducing pain and disability. It has been reported that progressive submaximal exercise program including cervicothoracic strengthening, endurance, flexibility, and coordination exercises has positive effects on chronic neck pain, related disability, quality of life and mood. In this study, in addition to telerehabilitation-based PNE, progressive submaximal exercise program will also be given to the participants through telerehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-55
* History of neck pain lasting at least three months
* Agreeing to participate in the study
* Being able to read and write Turkish
* Having a computer or tablet and an active internet connection at home
* To be able to use a computer, tablet and internet at a level to participate in video conference or to have a relative who can help in this regard.

Exclusion Criteria:

* History of spinal surgery
* Traumatic cervical injuries
* Serious comorbidities (neurological, neuromuscular, cardiological, psychiatric)
* Tumor conditions
* Having vision and hearing problems
* Cognitive problems
* Receiving physiotherapy for neck and/or low back pain in the last 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 6 weeks
  Numerical Pain Rating Scale will be used to evaluate the severity of pain. Participants will be asked to determine the number that best describes their pain, with 0 = no pain and 10 = unbearable pain, on a scale divided into numbers between 0 and 10 for the severity of pain they feel during rest and activity.
Neurophysiology of Pain Questionnaire | 6 weeks
  The Neurophysiology of Pain Questionnaire will be used to assess pain information. The Pain Neurophysiology Questionnaire was developed as a method of assessing whether healthcare professionals and patients understand the pain and its underlying complex neurophysiological mechanisms. Scoring is in the range of 0-13 points according to the number of correct answers given. Higher scores mean better pain knowledge. It is widely used by clinicians to monitor information exchange in pain education interventions.

SECONDARY OUTCOMES:
Neck Disability Index | 6 weeks
  The level of disability associated with the neck pain will be evaluated with the Neck Disability Index. The ındex consists of 10 sections that include pain sensitivity, personal care, weight lifting, reading, headaches, concentration, work/job, driving, sleep, and social activities. Each item is scored between zero (no disability) and five (total disability). The maximum score is therefore 50. Higher scores indicate having more disabilities.
Tampa Scale of Kinesiophobia | 6 weeks
  Tampa Kinesiophobia Scale will be used to evaluate kinesiophobia, which is an anxiety state that develops against activity and physical movement due to pain and fear of re-injury. The scale has 17 pain statements, and the patient selected her agreement for each question using a 4-point scale. The maximum score is 68. Higher score indicates having more fear of movement.
Pain Catastrophising Scale | 6 weeks
  Pain Catastrophising Scale will be used to determine the degree of pain catastrophising felt by individuals with pain. Pain Catastrophising Scale is a self-reported scale with 13 statements, where the patient ranks the affirmations between 0 "minimal" to 4 "very intense." The calculation of the final score is based on 3 subdomains of the scale and scores closer to 52 indicate worse results.
World Health Organization Quality of Life Scale-Short Form (WHOQOL-Bref) | 6 weeks
  The Turkish version of the World Health Organization Quality of Life Scale Short Form (WHOQOL-BREF) will be used to assess the quality of life. The scale consists of 4 quality of life domains: physical, psychological, social relations and environmental. It has 27 statements and the maximum score is 135. Higher score means higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yesim SALIK SENGUL, Assoc. Prof., Principal Investigator — Dokuz Eylul University
Locations (1):
- School of Physical Therapy and Rehabilitation, Dokuz Eylül University, Izmir, Turkey (Türkiye)